CLINICAL TRIAL: NCT00197561
Title: Partnership on Nutrition and HIV/AIDS Research in Tanzania: Exploratory Research Study on Selenium and HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Wafaie Fawzi, Harvard School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD43555
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections; Pregnancy Complications
Keywords: HIV; Selenium; Nutrition; Women; Pregnancy; Tanzania; Maternal and child health outcomes; HIV/AIDS; Pregnancy Outcome
MeSH Terms: conditions — HIV Infections; Pregnancy Complications; Acquired Immunodeficiency Syndrome | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selenium (Active Comparator): Selenium (200 ug as selenomethionine)
  Interventions: Dietary Supplement: Selenium
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Taken orally once per day from randomization through delivery and through the first 6 months after delivery.
  Arms: Placebo
Dietary Supplement: Selenium — 200 ug of selenomethionine taken orally once per day from randomization through delivery and for the first 6 months after delivery
  Arms: Selenium

SUMMARY:
The purpose of this study is to determine whether the oral administration of daily selenium supplements to HIV-1 positive pregnant women: enhances immune status and reduces the HIV-1 viral load at six months postpartum, reduces the risk of lower genital shedding of HIV-1 infected cells at 36 weeks of gestation, and reduces the risk of mastitis at six weeks postpartum, compared to placebo.

DETAILED DESCRIPTION:
We are recruiting pregnant women who are infected with HIV and assign them to receive selenium or placebo. All women will be given standard prenatal care, including nevirapine for the prevention of mother-to-child transmission and prenatal multivitamin supplements. We will examine the effect of the selenium supplements on intermediate outcomes predictive of the risks of transmission of HIV and to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 Infected women between 12 and 27 weeks of gestation

Exclusion Criteria:

* Women with clinical AIDS defined according to WHO Criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2003-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change in CD4 cell counts and viral load from baseline to six weeks and six months postpartum in HIV-1 positive women | Enrollment (12-27 wks gestation) to 6 months postpartum
Risk of lower genital shedding of HIV-1 infected cells at 36 wks gestation | At 36 wks gestation

SECONDARY OUTCOMES:
Risk of subclinical mastitis as defined by elevated sodium concentrations in breastmilk at 6 weeks postpartum | 6 weeks postpartum
Fetal death, premature delivery, and low birth weight | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W. Fawzi, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Muhimibili University College of Health Scienes, Upanga, Dar Es Salaaam, Tanzania

REFERENCES:
- [Result] Kupka R, Mugusi F, Aboud S, Hertzmark E, Spiegelman D, Fawzi WW. Effect of selenium supplements on hemoglobin concentration and morbidity among HIV-1-infected Tanzanian women. Clin Infect Dis. 2009 May 15;48(10):1475-8. doi: 10.1086/598334. PMID 19368503
- [Derived] Kupka R, Mugusi F, Aboud S, Msamanga GI, Finkelstein JL, Spiegelman D, Fawzi WW. Randomized, double-blind, placebo-controlled trial of selenium supplements among HIV-infected pregnant women in Tanzania: effects on maternal and child outcomes. Am J Clin Nutr. 2008 Jun;87(6):1802-8. doi: 10.1093/ajcn/87.6.1802. PMID 18541571